CLINICAL TRIAL: NCT03638986
Title: Prospektive Studie Zum Vergleich Der Beiden Validierten Deutschen Versionen Des "Tinnitus Functional Index" für Die Schweiz Und für Deutschland
Brief Title: Comparison of the Two Validated German Versions of the "Tinnitus Functional Index" for Switzerland and for Germany
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: TFI_GER
Record Dates: First submitted 2018-08-13; First posted 2018-08-20 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Swiss version first: This group will first complete the Swiss version and second the German version of the TFI
  Interventions: Other: No intervention planned
- German version first: This group will first complete the German version and second the Swiss version of the TFI
  Interventions: Other: No intervention planned

INTERVENTIONS:
Other: No intervention planned — No Intervention planned.

SUMMARY:
Tinnitus is defined as a perception of sound without any external sound source. Chronic tinnitus is a frequent condition that can affect the quality of life. The questionnaire "Tinnitus Functional Index (TFI)" promises to be the new gold standard in tinnitus evaluation. Due to the forward and backward translation of this questionnaire, there are two different German versions of TFI for Switzerland and Germany. Both German versions were validated. The aim of this study is to compare the two German versions of the TFI with each other and to recommend the better one for the further use in tinnitus evaluation for the German speaking population.

ELIGIBILITY:
Inclusion Criteria:

* Electronic given informed consent
* Older than 18 years
* Existing tinnitus
* Sufficient knowledge of the German language

Exclusion Criteria:

* Insufficient knowledge of the German language
* Impossibility to fulfill an online questionnaire due to cognitive or physical limitation
* No tinnitus
* Younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with tinnitus
Sampling Method: Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the TFI sumscore of both German versions | 20 minutes
  TFI sumscore ranges from 0 to 100

SECONDARY OUTCOMES:
Factor analysis of the two German TFI versions | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Peter, MD, Principal Investigator — Universityhospital Zurich, ENT Department
Locations (2):
- Universitätsmedizin Berlin, Tinnituszentrum der Charité, Berlin, Germany
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meikle MB, Henry JA, Griest SE, Stewart BJ, Abrams HB, McArdle R, Myers PJ, Newman CW, Sandridge S, Turk DC, Folmer RL, Frederick EJ, House JW, Jacobson GP, Kinney SE, Martin WH, Nagler SM, Reich GE, Searchfield G, Sweetow R, Vernon JA. The tinnitus functional index: development of a new clinical measure for chronic, intrusive tinnitus. Ear Hear. 2012 Mar-Apr;33(2):153-76. doi: 10.1097/AUD.0b013e31822f67c0. PMID 22156949
- [Background] Peter N, Kleinjung T, Jeker R, Meyer M, Klaghofer R, Weidt S. Tinnitus functional index: validation of the German version for Switzerland. Health Qual Life Outcomes. 2017 May 5;15(1):94. doi: 10.1186/s12955-017-0669-x. PMID 28476163
- [Background] Bruggemann P, Szczepek AJ, Kleinjung T, Ojo M, Mazurek B. [Validation of the German Version of Tinnitus Functional Index (TFI)]. Laryngorhinootologie. 2017 Sep;96(9):615-619. doi: 10.1055/s-0042-122342. Epub 2017 May 12. German. PMID 28499301